CLINICAL TRIAL: NCT05448820
Title: A Phase 1/2 Study of YH001 in Combination With Envafolimab With or Without Doxorubicin in Patients With Advanced or Metastatic Sarcoma
Brief Title: YH001 Plus Envafolimab With or Without Doxorubicin in Patients With Advanced or Metastatic Sarcoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tracon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YH001/KN035SAR101
Record Dates: First submitted 2022-06-28; First posted 2022-07-07 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Advanced Sarcoma; Metastatic Sarcoma; Soft Tissue Sarcoma
Keywords: Tracon; STS; LMS; DDLS; ASPS; envafolimab; YH001; CTLA-4; PD-L1; chondrosarcoma
MeSH Terms: conditions — Sarcoma; Diabetes Mellitus, Insulin-Dependent, 12; Chondrosarcoma | interventions — envafolimab; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- P1 Cohort 1A: Dose 1 YH001 + Dose 1 Envafolimab Q3WK (Experimental): Dose 1 of YH001 will be dosed in combination with Dose 1 Envafolimab every 3 weeks.
  Interventions: Drug: YH001; Drug: Envafolimab
- P1 Cohort 2A: Dose 2 YH001 + Dose 1 Envafolimab Q3WK (Experimental): Dose 1 of YH001 will be dosed in combination with Dose 1 Envafolimab every 3 weeks.
  Interventions: Drug: YH001; Drug: Envafolimab
- P1 Cohort 1B: Dose 1 YH001 + Dose 1 Envafolimab + Doxorubicin Q3WK (Experimental): Dose 1 of YH001 will be dosed in combination with Dose 1 of Envafolimab with Doxorubicin every 3 weeks.
  Interventions: Drug: YH001; Drug: Envafolimab; Drug: Doxorubicin
- P1 Cohort 2B: Dose 2 YH001 + Dose 1 Envafolimab + Doxorubicin Q3WK (Experimental): Dose 1 of YH001 will be dosed in combination with Dose 1 of Envafolimab with Doxorubicin every 3 weeks.
  Interventions: Drug: YH001; Drug: Envafolimab; Drug: Doxorubicin
- P2: Sarcoma Subtype 1 RP2D YH001 + Dose 1 Envafolimab Q3WK (Experimental): Recommended Phase 2 Dose of YH001 in combination with Dose 1 of Envafolimab every 3 weeks
  Interventions: Drug: YH001; Drug: Envafolimab
- P2: Sarcoma Subtype 2 RP2D YH001 + Dose 1 Envafolimab Q3WK (Experimental): Recommended Phase 2 Dose of YH001 in combination with Dose 1 of Envafolimab every 3 weeks
  Interventions: Drug: YH001; Drug: Envafolimab
- P2: Sarcoma Subtype 3 RP2D YH001 + Dose 1 Envafolimab + Doxorubicin Q3WK (Experimental): Recommended Phase 2 Dose of YH001 in combination with Dose 1 of Envafolimab every 3 weeks and Doxorubicin every 3 weeks for a maximum of 6 doses
  Interventions: Drug: YH001; Drug: Envafolimab; Drug: Doxorubicin
- P2: Sarcoma Subtype 4 RP2D YH001 + Dose 1 Envafolimab + Doxorubicin Q3WK (Experimental): Recommended Phase 2 Dose of YH001 in combination with Dose 1 of Envafolimab every 3 weeks and Doxorubicin every 3 weeks for a maximum of 6 doses
  Interventions: Drug: YH001; Drug: Envafolimab; Drug: Doxorubicin

INTERVENTIONS:
Drug: YH001 — Anti-CTLA4 antibody
Drug: Envafolimab — Anti-PD-L1 antibody
  Other Names: KN035
Drug: Doxorubicin — Anthracycline
  Arms: P1 Cohort 1B: Dose 1 YH001 + Dose 1 Envafolimab + Doxorubicin Q3WK; P1 Cohort 2B: Dose 2 YH001 + Dose 1 Envafolimab + Doxorubicin Q3WK; P2: Sarcoma Subtype 3 RP2D YH001 + Dose 1 Envafolimab + Doxorubicin Q3WK; P2: Sarcoma Subtype 4 RP2D YH001 + Dose 1 Envafolimab + Doxorubicin Q3WK

SUMMARY:
This is a multicenter, open label, Phase 1/2 study of YH001 initially given in combination with envafolimab, and then given in combination with envafolimab plus doxorubicin in patients with advanced or metastatic sarcoma, followed by Phase 2 cohorts of patients with select histologies of advanced or metastatic sarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed advanced or metastatic sarcoma patients without UPS or MFS who are refractory to or intolerant to standard treatments for their disease.
2. Histologically confirmed advanced or metastatic sarcoma patients without UPS or MFS who have not received any immune checkpoint inhibitors or doxorubicin, and with histology for which doxorubicin is considered a reasonable treatment option (for Cohort 1B, 2B and Expanded Cohort 1B and/or 2B)
3. Measurable disease by RECIST 1.1
4. Age ≥ 18 years
5. Adequate organ function
6. Left ventricular ejection fraction (LVEF) as measured by echo or multigated acquisition scan of > 50% (for patients to receive doxorubicin)
7. Willingness and ability to consent for self to participate in study
8. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
9. Men who are sterile or agree to use a condom with spermicide .
10. Women of non-child bearing potential due to surgical sterilization or medically-documented ovarian failure confirmed by medical history, or women of child bearing potential who test negative for pregnancy at time of enrollment and agree to use at least 2 acceptable methods of birth control

Exclusion Criteria:

1. Gastrointestinal stromal tumor (GIST) or desmoid tumors
2. Condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days prior to enrollment
3. Known allergy to any component of any study drug that the patient would receive if enrolled into this study
4. Prior T-cell or NK-cell therapy
5. Prior pericardial or mediastinal radiation (for patients to receive doxorubicin)
6. Acute coronary syndromes within 6 months of enrollment
7. Women who are pregnant or breast feeding
8. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Determine recommended phase 2 dose of YH001 in combination with Envafolimab | 8 months
  Evaluate safety and tolerability and determine the recommended Phase 2 dose (RP2D) of YH001 when given with envafolimab dosed SC every 3 weeks in patients with advanced or metastatic sarcoma who are refractory to or intolerant to other available therapies.
Phase 1: Determine recommended phase 2 dose of YH001 in combination with Envafolimab with Doxorubicin | 8 months
  Evaluate safety and tolerability and determine RP2D of YH001 in combination with envafolimab dosed SC every 3 weeks and doxorubicin dosed every three weeks in patients with advanced or metastatic sarcoma who have not received doxorubicin and are refractory to or intolerant to other available therapies.
Phase 2: Determine the objective response rate (ORR) of YH001 in combination with Envafolimab and Doxorubicin | 18 months
  Determine the ORR of envafolimab, YH001 and doxorubicin by RECIST 1.1 by investigator assessment in patients who have not received immune checkpoint inhibitors or doxorubicin with subtypes of advanced or metastatic soft tissue sarcoma.
Phase 2: Determine the objective response rate (ORR) of YH001 in combination with Envafolimab | 22 months
  Determine the ORR of envafolimab and YH001 by RECIST 1.1 by investigator in patients with subtypes of advanced or metastatic soft tissue sarcoma who have not received immune checkpoint inhibitors.

SECONDARY OUTCOMES:
Phase 1: YH001 concentrations | 8 months
  Determine YH001 trough concentration when given with envafolimab with or without doxorubicin.
Phase 1: Envafolimab concentrations | 8 months
  Determine envafolimab trough concentration when given with YH001 with or without doxorubicin.
Phase 1: Determine the Rate of YH001 Immunogenicity | 8 months
  Evaluate the formation of YH001 anti-drug antibodies (ADA).
Phase 1: Determine the Rate of Envafolimab Immunogenicity | 8 months
  Evaluate the formation of envafolimab anti-drug antibodies (ADA).
Phase 1: Assessment of antitumor activity | 8 months
  Assess objective response rate (ORR) of YH001 by investigator using RECIST 1.1 when combined with envafolimab or envafolimab/doxorubicin combination in patients with advanced or metastatic sarcoma.
Phase 2: Determine the disease control rate (DCR) | 22 months
  Determine the Disease Control Rate of envafolimab, YH001 and doxorubicin or envafolimab and YH001 in patients with advanced or metastatic sarcoma.
Phase 2: Determine duration of response (DOR) | 22 months
  Determine the Duration of Response of envafolimab, YH001 and doxorubicin or envafolimab and YH001 in patients with advanced or metastatic sarcoma.
Phase 2: Determine Progression Free Survival (PFS) | 22 months
  Determine Progression Free Survival of envafolimab, YH001 and doxorubicin or envafolimab and YH001 in patients with advanced or metastatic sarcoma.
Phase 2: Determine Overall Survival (OS) | 22 months
  Determine Overall Survival of envafolimab, YH001 and doxorubicin or envafolimab and YH001 in patients with advanced or metastatic sarcoma.
Phase 2: YH001 concentration | 22 months
  Determine YH001 trough concentration when given with envafolimab with or without doxorubicin.
Phase 2: Envafolimab concentration | 22 months
  Determine envafolimab trough concentration when given with YH001 with or without doxorubicin.
Phase 2: Determine the Rate of YH001 Immunogenicity | 22 months
  Evaluate the formation of YH001 anti-drug antibodies (ADA).
Phase 2: Determine the Rate of Envafolimab Immunogenicity | 22 months
  Evaluate the formation of envafolimab anti-drug antibodies (ADA).
Phase 2: Type Incidence and Severity of Adverse Events | 25 months
  Type, incidence, severity (graded by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] Version 5.0), timing, seriousness, and relatedness of AEs and laboratory abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: James Freddo, MD, Study Director — Medical Monitor
Locations (6):
- United States (6):
  - Sarcoma Oncology Center, Santa Monica, California
  - Northwestern University, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- See also: TRACON Pharmaceuticals — http://www.traconpharma.com